CLINICAL TRIAL: NCT05619250
Title: Efficacy and Cost-effectiveness of Supervised Center-based Versus Unsupervised Home-based Training Programs in Older Adults: the PRO-Training Randomized Controlled Trial
Brief Title: Supervised Center-based vs. Unsupervised Home-based Exercise Programs (PRO-Training)
Acronym: PRO-Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Biomedical Research Networking Center on Frailty and Healthy Aging (CIBERFES) (Unknown); Complejo Hospitalario de Toledo (Other)
Responsible Party: Principal Investigator, Asier Mañas Bote, Principal investigator, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC-CHTO-881
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Physical Inactivity; Healthy; Older Adult
Keywords: Aging; Exercise; Physical activity; Supervised; Center-based; Unsupervised; Home-based; App-based; mHealth; Mobile app; Multicomponent training; Physical health; Mental health; Quality of life; Physical function; Cost-effectiveness
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Unsupervised home-based exercise group without motivational intervention (UNSUP) (Experimental): Participants will use a mobile application to perform a home-based training program autonomously, without the face-to-face supervision of a specialist during its execution.
  Interventions: Behavioral: Unsupervised home-based exercise group without motivational intervention (UNSUP)
- Unsupervised home-based exercise group with motivational intervention (UNSUP+) (Experimental): Participants will use a mobile application to perform a home-based training program autonomously, without the face-to-face supervision of a specialist during its execution. As opposed to the "UNSUP" group, the "UNSUP+" group will receive a motivational intervention.
  Interventions: Behavioral: Unsupervised home-based exercise group with motivational intervention (UNSUP+)
- Supervised center-based exercise group without motivational intervention (SUP) (Experimental): Participants will perform a center-based training program in small groups with a maximum of 8 participants per session, being supervised by an exercise professional.
  Interventions: Behavioral: Supervised center-based exercise group without motivational intervention (SUP)
- Supervised center-based exercise group with motivational intervention (SUP+) (Experimental): Participants will perform a center-based training program in small groups with a maximum of 8 participants per session, being supervised by an exercise professional. As opposed to the "SUP" group, the "SUP+" group will receive a motivational intervention.
  Interventions: Behavioral: Supervised center-based exercise group with motivational intervention (SUP+)
- Control group (CON) (No Intervention): Participants will not perform any type of exercise program during the intervention period and will be advised to maintain their usual lifestyle.

INTERVENTIONS:
Behavioral: Unsupervised home-based exercise group without motivational intervention (UNSUP) — UNSUP will receive a non-supervised physical exercise intervention using a mobile app at home. The UNSUP training program comprises the same exercise structure and is based on the same muscle groups and movements as the supervised groups, but is adapted to be performed at home with the use of elastic bands and the participant's own body weight. The exercise program will be divided into 3 different levels. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks.
  Arms: Unsupervised home-based exercise group without motivational intervention (UNSUP)
Behavioral: Unsupervised home-based exercise group with motivational intervention (UNSUP+) — UNSUP+ will receive a non-supervised physical exercise intervention using a mobile app at home. The UNSUP+ training program comprises the same exercise structure and is based on the same muscle groups and movements as the supervised groups, but is adapted to be performed at home with the use of elastic bands and the participant's own body weight. The exercise program will be divided into 3 different levels. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks. Further, motivational strategies will be applied based on self-determination theory.
  Arms: Unsupervised home-based exercise group with motivational intervention (UNSUP+)
Behavioral: Supervised center-based exercise group without motivational intervention (SUP) — SUP will attend the university facilities and will perform training in small groups, being supervised by an exercise professional. The SUP training program comprises the same exercise structure and is based on the same muscle groups and movements as the unsupervised groups, but is performed in a center using the equipment available at the facility (weight machines, free weight, stationary bikes, etc.). The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises (for upper and lower limbs), 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks.
  Arms: Supervised center-based exercise group without motivational intervention (SUP)
Behavioral: Supervised center-based exercise group with motivational intervention (SUP+) — SUP+ will attend the university facilities and will perform training in small groups, being supervised by an exercise professional. The SUP+ training program comprises the same exercise structure and is based on the same muscle groups and movements as the unsupervised groups, but is performed in a center using the equipment available at the facility (weight machines, free weight, stationary bikes, etc.). The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises (for upper and lower limbs), 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks. Further, motivational strategies will be applied based on self-determination theory.
  Arms: Supervised center-based exercise group with motivational intervention (SUP+)

SUMMARY:
The superiority of supervised center-based training programs compared with unsupervised home-based ones in older adults remains unclear, and no evidence exists on whether including a motivational component could moderate these differences. The present randomized controlled trial aims to determine the role of supervision and motivational strategies on the safety, adherence, efficacy, and cost-effectiveness of different training programs for improving physical and mental health in older adults. Participants (n=120, aged 60-75 years old) will be randomly divided into five groups: 1- Control group, 2- Unsupervised home-based exercise group without motivational intervention (UNSUP), 3- Unsupervised home-based exercise group with motivational intervention (UNSUP+), 4- Supervised center-based exercise group without motivational intervention (SUP) and 5- Supervised center-based exercise group with motivational intervention (SUP+). Participants assigned to the exercise groups will participate in a 24-week multicomponent exercise program (3 sessions/week, 60 min/session), while participants in the control group will be asked to maintain their usual lifestyle. Physical and mental health outcomes will be assessed, including lower and upper-body muscular function, physical function, cardiorespiratory function, anthropometry and body composition, health-related quality of life, cognitive performance, anxiety and depression status, physical activity and sedentary behavior, sleep, biochemical markers, motivators and barriers to exercise, individual's psychological needs, and level of self-determination. Assessments will be conducted at baseline (week 0), mid-intervention (week 12), at the end of the intervention period (week 25), and 24 weeks after the exercise intervention (week 48).

DETAILED DESCRIPTION:
Life expectancy for the Spanish population has increased to 85 years for women and 79 years for men, and it is estimated that Spain will be the second oldest country in the world by 2050. This fact contains an inevitable economic and public health challenge. Physical exercise is an effective intervention to attenuate the aging-related decline in physical function and well-being as well as for reducing morbidity and mortality risk. Current guidelines on physical activity (PA) by the World Health Organization (WHO) recommend that older adults perform at least 150-300 min/week of moderate-intensity aerobic PA, 75-150 min/week of vigorous-intensity aerobic PA, or a combination of both, as well as at least 3 days of strength and balance exercise. However, a large part of the older adult population does not meet the general recommendations for PA. This could be at least partly due to the fact that this type of population may have some limitations when starting a supervised center-based physical training program. In this regard, evidence overall shows that supervised center-based training programs are usually limited by issues such as economic constraints, convenience, and access or time commitments. Moreover, there are unpopulated areas comprising a large percentage of older people without direct access to facilities and qualified professionals to engage in effective physical activity. Besides that, the COVID-19 pandemic has opened an opportunity to carry out training programs from home without the supervision of a professional. If effective and safe, these interventions would represent an alternative to increasing the accessibility of physical exercise for older adults.

To date, there is a lack of consensus on the effectiveness, safety, and adherence of unsupervised home-based training programs. Several investigations have shown greater effectiveness on different health variables in exercise programs conducted under the supervision of a professional compared to those performed autonomously at home. However, some studies suggest that a home-based exercise intervention could be as effective as a supervised one. Furthermore, meta-analytical evidence recently published by the research team of this project found that the adherence rate to unsupervised physical exercise programs was low, and the intensity applied was not adequately prescribed. It is important to note that the lack of motivation in unsupervised programs might play an important role in these findings. Thus, the use of motivational strategies that foster autonomous motivation might help increase adherence to unsupervised exercise programs, with this adherence being a key factor for achieving health adaptations.

Therefore, studies analyzing how to cover all these limitations of unsupervised physical exercise are warranted to answer this research question. Along these lines, an adequate prescription of exercise dose and the implementation of motivational techniques could compensate for the lack of physiological stimulus and low adherence typically observed with this type of training program. Furthermore, there is no evidence comparing the cost-effectiveness, safety, and adherence of supervised face-to-face intervention vs online supervised intervention with and without motivational strategies. Under this context, the aim of this randomized controlled trial (RCT) will be to determine the efficacy, cost-effectiveness, safety, and adherence of different exercise training programs with or without supervision and the inclusion of motivational techniques in older adults.

Participants (n= 120; men and women aged 60-75 years old) will be divided into 5 groups: 1- Control group, 2- Unsupervised home-based exercise group without motivational intervention (UNSUP), 3- Unsupervised home-based exercise group with motivational intervention (UNSUP+), 4- Supervised center-based exercise group without motivational intervention (SUP) and 5- Supervised center-based exercise group with motivational intervention (SUP+). Exercise groups will perform physical exercise 3 days a week (1-hour sessions) for 24 weeks, with these sessions being performed from home (with the help of a mobile application that will be developed for this purpose) or at a center with the direct supervision of an exercise professional, according to the assigned group. The primary outcome will be lower-body muscular function. Secondary outcomes will be upper-body muscular function, physical function, cardiorespiratory function, anthropometry and body composition, health-related quality of life, cognitive performance, anxiety and depression status, physical activity and sedentary behavior, sleep, biochemical markers, motivators and barriers to exercise, individual's psychological needs, and level of self-determination. Further, an analysis of the costs of the programs (cost-effectiveness and cost-utility), adherence (rate of adherence to the exercise program), and safety (falls and adverse events) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* People aged between 60 and 75 years old.
* Being able to speak and read fluent Spanish.
* Being able to walk independently.
* Being physically able to participate in an exercise program.
* Having a smartphone and being able to understand and use mobile applications autonomously.

Exclusion Criteria:

* Acute or terminal illness.
* Myocardial infarction, coronary artery bypass grafting, angioplasty, angina, or other cardiac condition in the past year.
* Uncontrolled medical problems that the general practitioner considers would preclude patients from undertaking the exercise program (e.g., acute systemic illness such as pneumonia, acute rheumatoid arthritis, and acute or unstable heart failure).
* Conditions requiring a specialized physical exercise program (e.g., uncontrolled epilepsy, significant neurological disease or impairment, inability to maintain an upright seated position or unable to move independently, multiple sclerosis, cancer, Parkinson's, Alzheimer's, or chronic obstructive pulmonary disease).
* General practitioner-diagnosed hypertension that has not been controlled.
* Type I Diabetes or uncontrolled Type II Diabetes.
* History of major psychiatric illness including schizophrenia, generalized anxiety disorder, or depression according to the DSM-5.
* Morbid obesity (body mass index >39)
* Three or more self-reported falls in the last year.
* Not living in the community (e.g., living in nursing homes).
* Having participated in an exercise program during the 6 months prior to the study.
* Diagnosis of COVID-19 with hospitalization in intensive care unit.
* Any other consideration that interferes with the study aims and could be a risk to the participant, at the discretion of the researcher and the general practitioner.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-07-19 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Lower-body muscular function | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  The force-velocity relationship and the rate of force development (RFD) will be assessed on a horizontal leg press device (Technogym, Element, Italy) instrumented with a force plate (Type 9286BA, Kistler, Switzerland) and a linear position transducer device (TForce System, Ergotech, Spain). A familiarization session will be performed in session one before the evaluation day in session number three.
Costs | Through intervention completion, that is 24 weeks.
  Researchers will calculate total costs and costs per participant for each of the intervention groups. Mean difference in quality-adjusted life-year (QALY) scores at the end of the intervention will be assessed to analyze the cost-utility. Furthermore, an incremental cost-effectiveness ratio (ICER) will be assessed. Data on health-related quality of life measured by EQ-5D will be used for the calculations.
Adherence to physical training program | Through study completion, that is 48 weeks.
  Adherence to physical training program will be recorded in the unsupervised training groups using the mobile app. Trainers will record adherence to physical training program in the supervised training groups. It will be calculated as a percentage ([sessions completed/total sessions expected] x 100), where 0 % indicates total non-adherence and 100 % indicates full adherence to the exercise prescription. During the 24-week follow-up, we will assess through an ad-hoc self-reported questionnaire whether or not participants exercised, the exercise modality performed (supervised center-based and/or unsupervised home-based), and the number of weekly exercise sessions performed. The questionnaire will be administered on a weekly basis in written form.
Falls and adverse events | Through intervention completion, that is 24 weeks.
  Participants in the unsupervised and control groups will record in a diary their falls and adverse events during and outside exercise sessions. In the supervised groups, supervisors will register the incidence of falls during exercise sessions and participants will register them outside the exercise sessions using the diary.

SECONDARY OUTCOMES:
Upper-body muscular function | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  Grip strength will be measured with a standard hydraulic hand-held dynamometer on both arms (Takei TKK5401, Tokyo, Japan).
Maximum walking speed (10-m) | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  Time the participant takes to walk 10 meters at maximum speed without running.
Usual walking speed (3, 6 and 10-m) | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  Time the participant spends walking 3, 6 and 10 meters at their usual pace.
Short Physical Performance Battery (SPPB) | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  To assess the ability to stand with feet together in side-to-side, semi-tandem, and tandem positions (balance), 4-meters walk test (speed), and 5 times sit-to-stand (muscle power).
Senior Fitness Test (SFT) | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  SFT battery includes 30-second chair stand test (lower-body strength), 30-second arm curl test (upper-body strength), 6-minute walk test (aerobic endurance), Chair sit-and-reach test (lower-body flexibility), Back scratch test (upper-body flexibility) and 8-foot up-and-go test (agility and dynamic balance).
Cardiorespiratory function | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Cardiorespiratory function will be assessed by a maximal incremental cycloergometer test using a gas analyzer (Cosmed QUARK, Italy). An electrocardiogram will be performed both at rest and during exercise to evaluate the electrical activity of the heart.
Blood pressure | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  Systolic and diastolic blood pressure and heart rate will be assessed at rest using a digital upper arm blood pressure monitor (OMRON M2, Spain).
Anthropometry | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  Height and body mass will be measured with a stadiometer and scale (Seca 711, Hamburg, Germany) without shoes to the nearest 0.1 cm and 0.1 kg, respectively, and body mass index will be calculated. In addition, the perimeters of the neck, waist, and hip will be measured.
Body composition | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Four bone densitometry tests will be performed on each subject (whole body, forearm, lumbar spine, and femoral neck) using bone densitometry (Hologic Series Horizon-A, Bedford, United States). For the determination of muscle, fat, and bone mass, the results of the whole-body test will be used. For regional analysis, values from all tests will be used.
Health-related quality of life | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  The EuroQol-5D questionnaire will be used for assessing the health status of the participants, including a descriptive system formed by five dimensions and a visual analogue scale.
Cognitive Performance | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  The Trail-Making Test Part A and B, the Montreal Cognitive Assessment (MoCA) and the Digital Symbol Substitution test will be administered in the cognitive evaluation.
Anxiety | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The Zung Anxiety Self-Assessment Scale will be used.
Depression | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The short form of the Yesavage Geriatric Depression Scale will be used.
Physical activity and sedentary behavior patterns | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Physical activity and sedentary behavior will be assessed by accelerometry (GeneActiv Original, Activinsights, UK). The devices will be placed on the subject's non-dominant wrist using a watch strap for 8 days.
Sleep | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The number of hours of sleep will be assessed by accelerometry (GeneActiv Original, Activinsights, UK). In addition, the Pittsburgh Sleep Quality Index will be used as an additional instrument.
Biochemical markers | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Blood samples will be collected at rest after an overnight fast (>12 h). Samples will be collected at least 72-96 h apart from any exercise or testing session. Samples will be analyzed immediately for routine clinical chemistry measurements and then, they will be put into 500-µL aliquots and frozen at -80ºC for later analysis.
Motivators and barriers to exercise | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Motivators and barriers to exercise will be measured using the Exercise Benefits/Barriers Scale.
Motivation to exercise according to self-determination theory | Baseline (week 0), mid-intervention (week 12), post-intervention (week 25), and follow-up (week 48).
  For the evaluation of motivation according to the self-determination theory, the Behavioral Regulation during Exercise Questionnaire (BREQ-3) will be used.
Basic Psychological Needs in Exercise | Post-intervention (week 25) and follow-up (week 48).
  The Basic Psychological Needs in Exercise Scale (BPNES) will be used to assess the satisfaction of the three needs autonomy, competence, and relatedness in the exercise domain.

CONTACTS AND LOCATIONS:
Overall Officials: Asier Mañas, Ph.D., Principal Investigator — GENUD Toledo Research Group, University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha, Toledo, Castilla-La Mancha/Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Redondo P, Alcazar J, Valenzuela PL, Ara I, Alegre LM, Manas A. Validity of repetitions in reserve for prescribing resistance exercise in older adults. Exp Gerontol. 2025 Oct 15;210:112884. doi: 10.1016/j.exger.2025.112884. Epub 2025 Sep 2. PMID 40902458
- [Derived] Leal-Martin J, Munoz-Munoz M, Sierra-Ramon M, Cerezo-Arroyo M, Gomez-Redondo P, Alegre LM, Ara I, Garcia-Garcia FJ, Manas A. Metabolic equivalents intensity thresholds for physical activity classification in older adults. Eur Rev Aging Phys Act. 2024 May 21;21(1):14. doi: 10.1186/s11556-024-00348-5. PMID 38773408
- [Derived] Gomez-Redondo P, Valenzuela PL, Martinez-de-Quel O, Sanchez-Martin C, Cerezo-Arroyo M, Moreno-Manzanaro D, Alegre LM, Guadalupe-Grau A, Ara I, Manas A. The role of supervision and motivation during exercise on physical and mental health in older adults: a study protocol for a randomized controlled trial (PRO-Training project). BMC Geriatr. 2024 Mar 20;24(1):274. doi: 10.1186/s12877-024-04868-8. PMID 38509514